CLINICAL TRIAL: NCT02527265
Title: Open-label, Single-arm, Multiple-dose Safety, Titration, and Pharmacokinetic Trial of Afrezza® in Pediatric Patients Ages 4 to 17 Years With Type 1 Diabetes Mellitus
Brief Title: Afrezza Safety and Pharmacokinetics Study in Pediatric Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mannkind Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MKC-TI-155 Part 1; U1111-1166-5528 (Other: UTN)
Record Dates: First submitted 2015-08-17; First posted 2015-08-18 (Estimated); Results first posted 2021-04-06 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-03

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Afrezza (Technosphere Insulin) (Experimental): Individualized dose of Afrezza (Technosphere Insulin) for each patient at each meal (breakfast, lunch, and dinner) for 30 days.
  During the trial, all patients will receive multiple injections of basal long acting insulin, in general at bedtime every day.
  Interventions: Biological: Afrezza

INTERVENTIONS:
Biological: Afrezza — Pharmaceutical form: powder
  Route of administration: inhalation
  Other Names: Technosphere Insulin

SUMMARY:
Primary Objective:

-To assess the safety and tolerability of Afrezza in children ages 4 to 17 years with type 1 diabetes mellitus (T1DM).

Secondary Objectives:

* To assess the ability to titrate the prandial and supplemental doses of Afrezza at each meal.
* To assess pharmacokinetics (PK) following a prandial dose of Afrezza in children ages 4 to 17 years with T1DM.

DETAILED DESCRIPTION:
The patients are expected to participate in the study for approximately 6 to 8 weeks from Screening to final follow-up visit.

ELIGIBILITY:
Inclusion criteria :

1. Written or oral assent from the pediatric subject and written informed consent from the parent(s) or legal guardian and a witness, as required by both state and federal laws and the local Institutional Review Board;
2. Children aged ≥4 and ≤17 years (enrolled sequentially into 3 age cohorts: 13 to 17, 8 to 12, and 4 to 7 years);
3. Clinical diagnosis of T1DM and using insulin for at least 1 year;
4. Currently receiving a regimen of basal/bolus insulin administered by MDI for at least 6 weeks prior to enrollment;
5. Subjects with pre-breakfast self monitored blood glucose values between 80 and 250 mg/dL for 5 of 7 documented daily readings obtained in the week prior to Visit 2 (readings to be taken using glucometer provided at Screening Visit 1) and reported via the e Diary;
6. Subjects on a regimen of insulin via continuous SC insulin infusion may be enrolled if they satisfy all other enrollment criteria and are willing to convert to MDI for the duration of the study, beginning 6 weeks prior to enrollment. They must continue to meet all enrollment criteria after converting to the MDI regimen;
7. Total daily insulin dose ≤1.5 units/kg/day with a minimum of 3 units of RAA at every meal.
8. Hemoglobin A1c (HbA1c) ≥7.0% to <10.0% at the time of screening;
9. Fasting serum C-peptide ≤0.3 ng/mL;
10. Forced expiratory volume in 1 second (FEV1) ≥70% of National Health and Nutrition Examination Survey (NHANES) III predicted for children ≥8 years of age or Wang predicted for children <8 years of age;
11. Forced vital capacity ≥70% of NHANES III predicted for children ≥8 years of age or Wang predicted for children <8 years of age;
12. Females of childbearing potential, must use "highly effective" methods of contraception throughout conduct of the trial

Exclusion criteria:

1. Body mass index below 25th or above 95th percentile for age and gender according to Centers for Disease Control and Prevention growth charts;
2. History of physician diagnosis of asthma or any other clinically important pulmonary disease, or use of any medications to treat such conditions within the last year;
3. Allergy or known hypersensitivity for AFREZZA or to drugs with similar chemical structure;
4. Unstable diabetes control, defined as 2 or more episodes of severe hypoglycemia (i.e., an episode associated with a seizure, coma, or loss of consciousness) or any hospitalization or emergency room visit for poor diabetes control, ketoacidosis, hypoglycemia, or hyperglycemia within the preceding 3 months from screening;
5. Serum creatinine ≥ the upper limit of normal for age;
6. Respiratory tract infection within 30 days before screening or between screening and initiation of treatment period; subject may return 4 weeks after resolution of the infection for rescreening;
7. Evidence of any complication of diabetes (proliferative retinopathy, autonomic neuropathy, nephropathy, etc), or likelihood of requiring laser photocoagulation, vitrectomy, or other specific treatment for diabetic retinopathy in the coming year;
8. Smoking of tobacco or other substances or positive urine cotinine testing (>100 ng/mL);
9. Positive urine drug screen;
10. Positive urine pregnancy test for female subjects of childbearing potential;
11. Inability to perform study procedures including pulmonary function testing;
12. Exposure to any investigational product(s) in the past 3 months or 5 half-lives, whichever is more;
13. History of eating disorder;
14. Any disease or exposure to any medication which, in the judgment of the principal Investigator, may impact glucose metabolism;
15. Any concurrent medical or major psychiatric condition that makes the subject unsuitable for the clinical study or impairs the subject's ability to participate in the study.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2017-09-28 (Actual); Primary Completion 2020-03-17 (Actual); Study Completion 2020-06-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Operations, Study Director — Mannkind Corporation
Locations (13):
- United States (13):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Barbara Davis Center for Childhood Diabetes, Aurora, Colorado
  - Yale University Hospital, New Haven, Connecticut
  - University of Florida, Gainesville, Florida
  - USF Diabetes Center, Tampa, Florida
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Van Meter Pediatric Endocrinology, P.C., Atlanta, Georgia
  - Emory University Children's Center, Atlanta, Georgia
  - Indiana University, Riley Hospital for Children, Indianapolis, Indiana
  - Barry J. Reiner, MD, LLC, Baltimore, Maryland
  - Diabetes, Obesity, Cardiovascular Clinical Specialists (DOCS), Las Vegas, Nevada
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Le Bonheur Children's Hospital, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Haller MJ, Jones MC, Bhavsar S, Kaiserman KB. Time-Action Profile of Technosphere Insulin in Children with Type 1 Diabetes. Diabetes Ther. 2023 Mar;14(3):611-617. doi: 10.1007/s13300-023-01368-7. Epub 2023 Jan 18. PMID 36652106

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 48 subjects were screened for the study, of which 30 subjects were enrolled in the study (15 subjects each in Cohort 1 and Cohort 2)
Groups:
- Afrezza Cohort 1 (Ages 13-17); Afrezza Cohort 2 (Ages 8-12): Individualized dose of Afrezza (Technosphere Insulin) for each patient at each meal (breakfast, lunch, and dinner) for 30 days.
  During the trial, all patients will receive daily injections of basal long acting insulin, in general at bedtime every day.
  Afrezza: Pharmaceutical form: powder
  Route of administration: inhalation
Period: Overall Study
Arm/Group | Afrezza Cohort 1 (Ages 13-17) | Afrezza Cohort 2 (Ages 8-12)
Started | 15 | 15
Completed | 13 | 11
Not Completed | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Afrezza Cohort 1 (Ages 13-17) | Afrezza Cohort 2 (Ages 8-12) | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.0 (1.73) | 10.4 (1.55) | 12.7 (2.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 18
  Male | 7 | 5 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 15 | 13 | 28
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 12 | 13 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Insulin Maximum Observed Concentration (Cmax)
Description: Insulin Cmax after a dose of Afrezza
Time Frame: 250 minutes post-dose
Population: All subjects without any major deviations related to study drug administration, and for whom any PK parameters are available, will be included in the PK population.
  Subjects who sneeze or cough right after AFREZZA inhalation for PK profiling will be considered as important deviations related to IMP and will be excluded for PK analysis.
Measure: Mean (Standard Deviation); unit: μU/mL
Groups:
- Afrezza Cohort 1 (Ages 13-17); Afrezza Cohort 2 (Ages 8-12): Individualized dose of Afrezza (Technosphere Insulin) for each patient at each meal (breakfast, lunch, and dinner) for 30 days.
  During the trial, all patients will receive multiple injections of basal long acting insulin, in general at bedtime every day.
  Afrezza: Pharmaceutical form: powder
  Route of administration: inhalation
Arm/Group | Afrezza Cohort 1 (Ages 13-17) | Afrezza Cohort 2 (Ages 8-12)
Number analyzed (Participants) | 15 | 13
μU/mL
  4 unit cartridge: number analyzed (Participants) | 2 | 4
  4 unit cartridge | 28.5 (5.77) | 102 (31.4)
  8 unit cartridge: number analyzed (Participants) | 6 | 8
  8 unit cartridge | 101 (42.1) | 133 (91.0)
  12 unit cartridge: number analyzed (Participants) | 6 | 1
  12 unit cartridge | 201 (118) | 251 (NA) — n=1
  16 unit cartridge: number analyzed (Participants) | 1 | 0
  16 unit cartridge | 105 (NA) — n=1 |

2. Secondary Outcome: Insulin Time to Reach Cmax (Tmax)
Description: Insulin Tmax after a dose of Afrezza
Time Frame: 250 minutes post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Afrezza Cohort 1 (Ages 13-17) | Afrezza Cohort 2 (Ages 8-12)
Number analyzed (Participants) | 15 | 13
minutes
  4 unit cartridge: number analyzed (Participants) | 2 | 4
  4 unit cartridge | 12.5 (3.54) | 9.5 (4.04)
  8 unit cartridge: number analyzed (Participants) | 6 | 8
  8 unit cartridge | 13.5 (5.47) | 14.1 (5.44)
  12 unit cartridge: number analyzed (Participants) | 6 | 1
  12 unit cartridge | 15.3 (3.27) | 10.0 (NA) — n=1
  16 unit cartridge: number analyzed (Participants) | 1 | 0
  16 unit cartridge | 20.0 (NA) — n=1 |

3. Secondary Outcome: Insulin Area Under Concentration Time Curve (AUC)
Description: Insulin AUC after a dose of Afrezza
Time Frame: 250 minutes post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: min*μU/mL
Arm/Group | Afrezza Cohort 1 (Ages 13-17) | Afrezza Cohort 2 (Ages 8-12)
Number analyzed (Participants) | 15 | 13
min*μU/mL
  4 unit cartridge: number analyzed (Participants) | 2 | 4
  4 unit cartridge | 1468 (1272) | 2931 (1011)
  8 unit cartridge: number analyzed (Participants) | 6 | 8
  8 unit cartridge | 4488 (2644) | 4975 (2921)
  12 unit cartridge: number analyzed (Participants) | 6 | 1
  12 unit cartridge | 6400 (3009) | 5971 (NA) — n=1
  16 unit cartridge: number analyzed (Participants) | 1 | 0
  16 unit cartridge | 5778 (NA) — n=1 |

4. Secondary Outcome: Assessment of Fumaryl Diketopiperazine (FDKP) Elimination Half-life (t1/2)
Description: FDKP (inert carrier excipient) calculated half life t1/2
Time Frame: Using PK data collected over 250 minutes post-dose of Afrezza
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Afrezza Cohort 1 (Ages 13-17) | Afrezza Cohort 2 (Ages 8-12)
Number analyzed (Participants) | 15 | 13
minutes
  4 unit cartridge: number analyzed (Participants) | 2 | 4
  4 unit cartridge | 103 (23.0) | 86.8 (6.35)
  8 unit cartridge: number analyzed (Participants) | 6 | 8
  8 unit cartridge | 123 (31.3) | 86.5 (15.8)
  12 unit cartridge: number analyzed (Participants) | 6 | 1
  12 unit cartridge | 109 (25.9) | 95.5 (NA) — n=1
  16 unit cartridge: number analyzed (Participants) | 1 | 0
  16 unit cartridge | 144 (NA) — n=1 |

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Afrezza Cohort 1 (Ages 13-17) | Afrezza Cohort 2 (Ages 8-12)
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 1/15 | 1/15
Other Adverse Events (participants affected / at risk) | 12/15 | 11/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Afrezza Cohort 1 (Ages 13-17) (N=15) | Afrezza Cohort 2 (Ages 8-12) (N=15)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Afrezza Cohort 1 (Ages 13-17) (N=15) | Afrezza Cohort 2 (Ages 8-12) (N=15)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 5 (5)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 3 (3)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1)
Tenderness (General disorders) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 0 (0) | 1 (1)
Urine cotinine test positive (Investigations) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dysmenorrhea (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 10 (48) | 10 (45)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-02-14): https://cdn.clinicaltrials.gov/large-docs/65/NCT02527265/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-17): https://cdn.clinicaltrials.gov/large-docs/65/NCT02527265/SAP_002.pdf